CLINICAL TRIAL: NCT05228600
Title: A Multi-Center, Open-Label, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of YL-13027 in Patients With Advanced Solid Tumors
Brief Title: YL-13027 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Collaborators: Yingli Pharma US, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL-13027-003
Record Dates: First submitted 2021-12-20; First posted 2022-02-08 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- YL-13027 (Experimental): YL-13027 is a novel small molecule TGF-βR1 inhibitor. 1.1.1. Chemical Properties
  Chemical Name:
  6-(5-fluoro-2-(6-methylpyridin-2-yl)phenyl)imidazo[1,2-a]pyridine-3-carboxamide Molecular Formula C20H15FN4O Molecular Weight 346.36 Formulation YL-13027 is provided as pink film coated tablets for oral administration in two strengths, 30 mg and 120 mg.
  Packaging and Storage YL-13027 tablets are packaged (30 tablets/bottle) in the 45 mL opaque HDPE bottles with child resistant polypropylene caps, induction-sealed inner polypropylene liners. YL-13027 tablets should be protected from light in a closed container and stored at room temperature.
  Stability The shelf-life of YL-13027 oral tablets is tentatively set at 24 months when stored at room temperature.
  Interventions: Drug: YL-13027

INTERVENTIONS:
Drug: YL-13027 — YL-13027 is a novel small molecule TGF-βR1 inhibitor. 1.1.1. Chemical Properties
  Chemical Name:
  6-(5-fluoro-2-(6-methylpyridin-2-yl)phenyl)imidazo[1,2-a]pyridine-3-carboxamide Molecular Formula C20H15FN4O Molecular Weight 346.36 Formulation YL-13027 is provided as pink film coated tablets for oral administration in two strengths, 30 mg and 120 mg.
  Packaging and Storage YL-13027 tablets are packaged (30 tablets/bottle) in the 45 mL opaque HDPE bottles with child resistant polypropylene caps, induction-sealed inner polypropylene liners. YL-13027 tablets should be protected from light in a closed container and stored at room temperature.
  Stability The shelf-life of YL-13027 oral tablets is tentatively set at 24 months when stored at room temperature.

SUMMARY:
Part 1 (Phase Ia):

This is a dose escalation, 3 + 3 design study, to evaluate the safety and tolerability, and to determine the RP2D of YL-13027 when administered b.i.d. in patients with advanced solid tumors. Up to 4 cohorts of 3-6 patients each will be treated in part 1 of the study. One cycle is 28 days.

Part 2:

This is a dose expansion phase to further evaluate the safety, tolerability and preliminary anti-tumor activity of YL-13027 at the RP2D.

DETAILED DESCRIPTION:
3.1.3. Parts 1 and 2: Patients will receive study treatment until criteria for study termination are met.

A Safety Follow-up Visit will be conducted 30 days (±7 days) after the last dose of study treatment Patients who discontinue study treatment for reasons other than disease progression will have post-treatment follow-up for disease assessment until start of new anticancer treatment, patient withdraws consent, is lost to follow-up, death, or until the Sponsor stops the study, whichever comes first.

Adverse events will be assessed using the NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.

Tumor response will be assessed by physical examination, computed tomography (CT) and/or magnetic resonance imaging (MRI) scan using RECIST 1.1 criteria, assessed by the investigator. Patients who discontinue study treatment for reasons other than disease progression will have post-treatment follow-up for disease assessment until start of new anticancer treatment, patient withdraws consent, is lost to follow-up, death, or until the Sponsor stops the study, whichever comes first.

Specific procedures to be performed during the study, as well as their prescribed times and associated visit windows, are outlined in the Schedule of Activities (SoA) see Appendix 1. Details of each procedure are provided in Section 7. The Safety Monitoring Committee (SMC) will monitor safety during the duration of the study. The SMC will make reviews based on Investigator site dose adjustments, adverse events, serious adverse events or discontinuation study treatment and make any appropriate recommendations to the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

-

In order to be eligible for participation in this trial, the patient must meet all the following inclusion criteria:

1. Patients with advanced solid tumors that is unresectable or metastatic and considered refractory to or not candidates for all available approved therapy.
2. Measurable disease with at least one lesion amenable to response assessment per RECIST 1.1.
3. Demonstrate adequate organ function as defined below. All screening laboratories should be performed within 7 days of study treatment initiation.

   System Laboratory Value Hematological Absolute neutrophil count (ANC)
   * 1.5 × 109/L Platelets
   * 100 × 109/L Hemoglobin
   * 9 g/dL or ≥5.6 mmol/L Renal Creatinine* or

     ≤1.5 × the upper limit of normal (ULN) or Measured or calculated creatinine clearance (CrCl) (Cockroft-Gault)
   * 50 mL/min for patient with creatinine levels >1.5 × institutional ULN Hepatic Total bilirubin

     * 1.5 × ULN or direct bilirubin ≤ULN for patients with total bilirubin levels > 1.5× ULN Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)
     * 2.5 × ULN or ≤5 × ULN for patients with liver metastases Cardiac CK-MB, Troponin T, BNP < ULN
4. Has a ECOG performance status of 0-1.
5. Life expectancy >12 weeks at baseline.
6. Women of childbearing potential must have negative serum or urine pregnancy test within 72 hours prior to receiving the first study drug administration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
7. For women of childbearing potential, must be willing to use an adequate method of contraception from 30 days prior to the first study drug administration and at least 3 months following last day study drug administration.
8. Male patients of childbearing potential must be surgically sterile, or must agree to use adequate method of contraception during the study and at least 3 months following the last day of study drug administration.
9. Age ≥18 years at screening.
10. Able and willing to provide written informed consent and to follow study instructions.
11. Washout from prior anti-tumor therapy:

Previous Treatment Length of Time Prior to (Study entry/enrollment/first dose of study treatment) Cytotoxic therapies

* 4 weeks Mitomycin C or nitrosoureas
* 6 weeks Small molecule inhibitors
* 2 weeks or 5x T1/2, whichever is longer Biologic agents (e.g., antibodies)
* 4weeks Immunotherapy (e.g., CTLA4, PD-1, PD-L1 inhibitors)
* 4 weeks Radiotherapy
* 4 weeks Limited field radiotherapy or palliative radiotherapy
* 2 weeks Major surgery, excluding biopsy
* 4 weeks. Patients with recent major surgery must have recovered, in the opinion of the investigator, from the toxicity and/or complication from the intervention before starting therapy

Exclusion Criteria:

* The patient will be excluded from participating in the trial if any of the following exclusion criteria are met:

  1. Prior therapy with a TGF-ß signaling targeted agent.
  2. Known symptomatic brain metastases requiring steroids above physiologic replacement doses.
  3. Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment.
  4. Live vaccines within 30 days of study treatment.
  5. Unresolved toxicities from prior therapy, defined as having not resolved to NCI CTCAE v.5.0 Grade ≤1 or baseline, with exception of endocrinopathies from prior therapy and successfully treated (such as hypothyroidism), alopecia, vitiligo, and ≤ grade 2 peripheral neuropathy.
  6. Human immunodeficiency virus (HIV) infection with a current or a known history of AIDS-defining illness or HIV infection with a CD4+ T cell count <350 cells/μL and an HIV viral load more than 400 copies/μL.
  7. Patients with active viral (any etiology) hepatitis are excluded. However, patients with serologic evidence of chronic hepatitis B virus (HBV) infection (defined by a positive hepatitis B surface antigen test and a positive anti-hepatitis core antigen antibody test) who have a viral load below the limit quantification (HBV DNA titer <1000 cps/mL or 200 IU/mL), and are not currently on viral suppressive therapy may be eligible and should be discussed with the Medical Monitor. Patients with a history of hepatitis C virus (HCV) infection who have completed curative antiviral treatment and have a viral load below the limit of quantitation may be eligible and should be discussed with the Medical Monitor.
  8. Any of the following cardiac criteria experienced currently or within the last 6 months:

     1. Congestive heart failure (New York Heart Association ≥ Class 2).
     2. Any clinically significant abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting electrocardiograms (ECGs), e.g., complete left bundle branch block or third-degree heart block.
     3. Acute coronary syndrome within 6 months.
     4. Clinically significant cardiac arrhythmia.
     5. Mean QTC interval corrected (Frederica) for heart rate >470 ms.
     6. Left ventricular ejection fraction (LVEF) <50% or the lower limit of normal (per institutional standard).
  9. Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses, or active infection, as determined by the investigator.
  10. Any condition that impairs a patient's ability to swallow whole pills. Presence of an active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of YL-13027, as determined by the investigator.
  11. History of interstitial lung disease.
  12. An active additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
  13. Known allergy to any component of YL-13027.
  14. Participation in another clinical trial of an investigational agent within 30 days of screening.
  15. Patient has known psychiatric, substance abuse or other disorders that would interfere with cooperation with the requirements of the trial, in the opinion of the investigator.
  16. Patients who are pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the screening visit through 3 months after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Frequency, duration and severity of Adverse Events and Serious Adverse Events | Throughout the study for approximately 2 years
  Primary Outcome Measure(s):
  Part 1:
  Frequency, duration and severity of Adverse Events and Serious Adverse Events.
  Part 2:
  Frequency, duration and severity of Adverse Events and Serious Adverse Events.

SECONDARY OUTCOMES:
Pharmacokinetics | Throughout the study for approximately 2 years
  Secondary Outcome Measures:
  • Pharmacokinetics of YL-13027; to include: AUC, AUClast, AUCinf, AUMC, Cmin, Cmax, CL, T1/2, Tmax, and Vd
ORR | Throughout the study for approximately 2 years
  Efficacy
  - Overall Response Rate (ORR).
DOR | Throughout the study for approximately 2 years
  • Efficacy
  - Duration of Response (DOR).
PFS | Throughout the study for approximately 2 years
  Efficacy
  - Progression Free Survival (PFS).
Duration of Stable Disease | Throughout the study for approximately 2 years
  Efficacy
  - Duration of Stable Disease
Clinical Benefit Rate | Throughout the study for approximately 2 years
  Efficacy
  - Clinical Benefit Rate (CR+PR+SD)

OTHER OUTCOMES:
Plasma tumor antigens | Throughout the study for approximately 2 years
  Exploratory Outcome Measures:
  • Plasma tumor antigens (as appropriate to cancer type, e.g., CA19-9, CEA) and biomarkers of TGF-ß signaling.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Ah Rodon, Ph D, Principal Investigator — MD Anderson Cancer Center Houston TX 77030; Trisha Wi Draper, Ph D, Principal Investigator — University of Cincinnati Cincinnati, OH 45267-0562; Martin E Gutierrez, MD, Principal Investigator — Hackensack University Medical Center Hackensack, NJ 07601; Ignacio Ga Laguna,, MD, Ph.D, Principal Investigator — Huntsman Cancer Institute Salt Lake City, UT 84112
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States